CLINICAL TRIAL: NCT04189926
Title: Physical Activity, Sedentary Behavior and Weight Status in Early Childhood
Brief Title: Linking Activity, Nutrition, and Child Health
Acronym: LAUNCH
Status: Completed | Type: Observational
Sponsor: University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Russell Pate, Professor, University of South Carolina
Other Study IDs: Pro00069562; R01HD091483 (NIH)
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Child Obesity
Keywords: Obesity; Physical Activity; Young Children; Sedentary Behavior; Childcare Centers; Family
MeSH Terms: conditions — Obesity; Pediatric Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Leading health organizations have identified prevention of obesity in young children as a critical public health challenge. Low levels of physical activity and high levels of sedentary behavior may contribute to the development of excessive fatness in young children, but these relationships have not been fully explored, and accelerometry rarely has been used to measure physical activity levels in infants and toddlers. No previous study has used accelerometry as an objective measure of physical activity in young children as they develop from infancy to preschool age. Accordingly, little is known about the factors associated with the development of physical activity behavior in very young children, and little is known about the influence of physical activity and sedentary behavior, measured objectively, on development of weight status during the transition from infancy to age 3. The first aim of this study is to describe physical activity and sedentary behavior in young children as they develop from infancy to preschool age. The second aim is to describe the longitudinal associations of weight status with physical activity and sedentary behavior as young children develop from infancy to preschool age. The proposed investigation will employ a longitudinal, observational study design. Participants will be 160 children and their biological mothers living in Columbia, South Carolina. For each participating child, measurements will be taken at 6, 12, 18, 24, 30, and 36 months of age. At each time point, each child's physical activity, sedentary behavior, weight status and motor developmental status will be measured objectively, and each child's mother will complete a survey to assess demographic, social and physical environmental factors; gross motor milestones; parenting practices related to physical activity and sedentary behavior; and dietary practices. Childcare center directors will complete a survey annually to assess center characteristics, and the Environment and Policy Assessment and Observation (EPAO) will be administered in the child's classroom annually.

DETAILED DESCRIPTION:
Subjects and Settings. The proposed research will be conducted in Columbia/Richland County, South Carolina (SC). Participants will be 160 children and their biological mothers. Children of all races and ethnic backgrounds will be included. Our recruitment procedures will be designed to produce a sample with the following approximate race/ethnicity distribution: 38% non-Hispanic African American, 38% non-Hispanic White, 20% Hispanic, and 4% other. Further, we anticipate that approximately two-thirds of the participating children be attending formal childcare centers and one-third will be at home or staying with a family member. Equal percentages of female and male children will be included. Children will be excluded from the study if they were born before 37 weeks gestation or have a physical limitation that would invalidate accelerometry as a measure of physical activity.

Recruitment of Participants. Participants in the study will be 160 mother-child dyads who will be recruited into the study when the children are between 3 and 6 months of age. They will be residents of Richland County, South Carolina. Recruitment will take place across a 9-month period and will be designed to recruit two cohorts of 80 children each. Baseline data collection will occur when each child is within one month of being 6 months of age. The recruitment process will be coordinated by Richland County First Steps (RCFS), a non-profit organization founded in 1999 to support provision of quality early childhood education for children ages 0 to 5 in Richland County.

One-third of participants will be mother-child dyads from families in which the child does not attend a formal childcare center. Richland County First Steps, in addition to its work with childcare centers, delivers programs directly to families of young children, including Latino families.

Cohort Maintenance. Participating mothers and children will be retained in the study across a 30-month period of observation by maintaining excellent communication with the parents and, for children attending formal childcare centers, the directors and staff of the childcare centers they attend. The process of maintaining excellent relationships with parents and center staff will be coordinated by RCFS and managed collaboratively with the University-based study staff.

Measures

Physical Activity and Sedentary Behavior. Total day physical activity and sedentary behavior will be measured objectively using an ActiGraph accelerometer (GT3X-BT model, Pensacola, FL). Accelerometers will be initialized prior to data collection and will be set to begin collecting data at midnight of the day of distribution. Children will be fitted with the accelerometer during a data collection visit with the parent and child at his/her childcare center, home or other appropriate location. Based on preliminary work, we anticipate creating two variables to define physical activity. The first variable will be based on counts per minute averaged across 7 days of wear. This expression of the data will be applicable to the full age range since intensity cutpoints have not been established for non-ambulatory children. The second expression will use age-specific cutpoints to determine minutes per hour of total physical activity and sedentary behavior.

Dietary Behavior. We will examine how diet, physical activity and sedentary behavior interact in influencing developmental trajectories for weight status in children transitioning from infancy to early childhood. Five instruments will be used in assessing children's dietary behavior. At baseline data collection (child age = 6 months) the mother will be asked to complete the Baby Eating Behavior Questionnaire 80, which will provide information on the child's appetite during the first three months of life, and the ECLS-B Parent Questionnaire (9-month version),81 which will provide information on the child's current and previous feeding behavior, including breast-feeding history. At subsequent data collection points (child age = 12 to 36 months) the mother will complete the ECLS-B Parent Questionnaire (24-month version), which will provide information on specific dietary behaviors, and the Multiple Indicator Cluster Survey (MICS) Dietary Intake survey, which will provide information on foods consumed by the child on the previous day. In addition, at the 18-month and 36-month data collection points, mothers will complete the Dietary Food Frequency Self-Administered Questionnaire as developed for use in the National Children's Study.

Sleep characteristics. Sleep behavior will be assessed via actigraphy in children whose parents consent to participation in this component of the protocol. Due to the substantial participant burden, participation in this procedure will be optional. All parents participating in the overall study will be invited to take part, and those who consent will receive an additional incentive. Participating children will wear an actigraph (MicroMini-Motionlogger, Ambulatory Monitoring, Inc.) 24 hours per day for seven days, except during bathing or other water activities.

Weight Status. At each timepoint, data collectors will measure weight and length/height using standard protocols. Age- and sex-specific weight-for-length percentiles and Z-scores will be calculated from weight and length according to the World Health Organization (WHO) growth charts. For children 24 months of age and older, the age- and sex-specific body mass index (BMI) percentiles and Z-scores will be calculated according to the CDC growth charts.

Demographic Characteristics. At the first measurement point, each child's biological mother will report her child's date of birth, gender, race/ethnicity, birth weight, length at birth, and gestational age. The mother will report her own age, race/ethnicity, marital status, and highest level of education achieved, which will be used as an indicator of socioeconomic status. The mother will also report information related to her pregnancy with the participating child.

Social Environmental Factors. At each measurement point, each child's mother will report her employment status, physical activity behavior, and screen media use. Mothers will report the number of other children living in the child's home and the age and gender of the children. Mothers will also report whether there is another adult that lives with the child. Mothers will also report the amount of time they spend playing with their child and the amount of time the child spends playing with children of a similar age.

Physical Environmental Factors. Each child's mother will report her child's sleep habits, outdoor play, television and screen media use, time spent in confining equipment, and care arrangements during weekdays. Mothers will also report physical activity equipment in the home. This information will be collected at each of the six time points.

Childcare Center Characteristics. For children attending childcare, we will conduct assessments of their center once per year. The goal will be to perform a comprehensive evaluation of the center's policies and practices related to nutrition and physical activity. Center directors will provide information about their center's characteristics and policies, and teachers will complete a survey about classroom practices related to physical activity and nutrition. The director survey will address global policies related to physical activity and nutrition as well as institutional characteristics. The teacher survey will address classroom practices, including physical activity, sedentary behavior, meals and snacks, and teacher behavior and engagement, using the Go NAP SACC self-assessment instrument.91 In addition, we will conduct observations of the childcare environment using the Environment and Policy Assessment and Observations (EPAO).92 The EPAO is a standardized instrument that has been used widely to assess physical activity and nutrition in childcare environments. The EPAO is completed by a trained observer during a full-day visit to a childcare center, during which a single classroom is observed. Scores on 8 nutrition and 8 physical activity subscales will be calculated as well as a total physical activity and total nutrition score for each center.

Motor Developmental Status. Each child's biological mother will report the age (in months) when her child first rolled over, sat unassisted, and began walking independently. In addition, motor developmental status will be assessed using the Peabody Developmental Motor Scales-2 (PDMS-2).94 Two trained data collectors will administer and score the PDMS-2; data collection will take place at the participating child's childcare center or other appropriate community location. The following gross movement subtests will be administered according to standard age-specific protocols: reflexes, stationary performances, locomotion and object manipulation. A Gross Motor Quotient will be calculated as the sum of the child's scores on three subtests. For children less than 1 year of age the sub-tests will be Reflexes, Stationary and Locomotion. For children ages 1 to 3 years the sub-tests will be Stationary, Locomotion, and Object Manipulation. Performance is reported as both a raw score and as an age-specific percentile.

Measurement Logistics. A total of 160 children, organized in two waves of 80 children each, will be measured. For each participating child, there will be six measurement time points at 6-, 12-, 18-, 24-, 30-, and 36-months of age, with data collection occurring +/- 1 month of the specified age. The same measurement protocol will be applied at each measurement time point. Each child will be assessed during two visits at each measurement time point. The first visit will include anthropometric measures, accelerometer distribution, and parent survey administration, and the second visit will include the motor development assessment. The first visit will take place at the child's home, at the childcare center or at another appropriate community location. The motor development assessment will take place at the childcare center or other appropriate community location. The motor development assessment will occur within two weeks of the first visit, but not during the week of accelerometer wear. All data collection procedures will be administered by trained and experienced research staff.

For children attending a childcare center, center directors will complete a survey annually to assess center characteristics. The classroom teacher(s) of participating children will complete a survey annually. The EPAO will be completed on each classroom serving a participating child once per year, or as children change to new classrooms. The EPAO will be completed by trained data collectors. The Measurement Coordinator will download data from the accelerometers as the monitors are collected, and the data will be scanned by the data collection staff on a weekly basis. Surveys, anthropometric forms, and observation forms will be entered into secure databases on a weekly basis. This measurement logistics plan is similar to the plan that has been used by this research team in two previous studies of physical activity in preschool children.

All data collected and entered will be reviewed weekly by the Measurement Coordinator for quality control of data entry and completeness. Quality control and data completeness reports will be generated monthly and discussed at project meetings. Reliability assessments of anthropometry and motor development assessments will be conducted at least twice per year for each data collector. Quality control visits will be conducted at least twice per year to participating childcare centers for the purpose of observing data collectors.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 6-36 months and their biological mothers, recruited from childcare centers and families in the greater Columbia, SC area

Exclusion Criteria:

* Children born prior to 37 weeks gestation or who have a physical limitation that would invalidate accelerometry as a measure of physical activity

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The proposed research will be conducted in Columbia/Richland County, South Carolina (SC). Participants will be 160 children and their biological mothers. Children of all races and ethnic backgrounds will be included. Our recruitment procedures will be designed to produce a sample with the following approximate race/ethnicity distribution: 38% non-Hispanic African American, 38% non-Hispanic White, 20% Hispanic, and 4% other. Further, we anticipate that approximately two-thirds of the participating children be attending formal childcare centers and one-third will be at home or staying with a family member. Equal percentages of female and male children will be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Total daily physical activity | Every 6 months, ages 6-36 months
  Average accelerometer counts per minute
Total physical activity | Every 6 months, ages 6-36 months
  Average accelerometer counts per minute above the light PA cutpoint
Sedentary behavior | Every 6 months, ages 6-36 months
  Average accelerometer counts per minute below the light PA cutpoint
Weight status | Every 6 months, ages 6-36 months
  Weight in kg
Dietary behavior | Every 6 months, ages 6-36 months
  ECLS-B and other parent report instruments
Sleep | Every 6 months, ages 6-36 months
  Sleep behavior measured by actigraph, measured in 50% of participants

CONTACTS AND LOCATIONS:
Overall Officials: Russell R Pate, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No